CLINICAL TRIAL: NCT04766957
Title: Pilot Clinical Trial on the Efficacy and Safety of IDRACARE® in Moderate to Severe Symptoms of Vulvovaginal Atrophy
Brief Title: Pilot Clinical Trial of IDRACARE® in Moderate to Severe Symptoms of Vulvovaginal Atrophy
Acronym: IDRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procare Health Iberia S.L. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IDRA
Record Dates: First submitted 2021-02-13; First posted 2021-02-23 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2022-12

CONDITIONS: Vulvovaginal Atrophy

STUDY DESIGN:
Intervention Model Description: open study, only one arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Idracare (Experimental): The treatment will be applied 2 times a week, preferably at night before going to bed.
  Interventions: Device: Idracare

INTERVENTIONS:
Device: Idracare — Treatment will last 3 months (12 weeks). The treatment will be applied 2 times a week, preferably at night before going to bed.

SUMMARY:
Pilot clinical trial on the efficacy and safety of IDRACARE® in moderate to severe symptoms of vulvovaginal atrophy. To assess the efficacy and safety of Idracare® in the treatment of symptoms of AVV (dryness and / or dyspareunia) associated with menopause.

DETAILED DESCRIPTION:
Pilot clinical trial on the efficacy and safety of IDRACARE® in moderate to severe symptoms of vulvovaginal atrophy. To assess the efficacy and safety of Idracare® in the treatment of symptoms of AVV (dryness and / or dyspareunia) associated with menopause.

Open study with only one arm. The study has a total duration per patient of 3 months: initial visit (V1), a follow-up visit (V2) after 4 weeks of treatment and a final visit (V3) after 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women who attend medical centers, either for a visit related to vulvovaginal atrophy (VVA) or for any other reason for consultation, with symptoms of VVA (dryness and / or dyspareunia) of moderate or severe intensity (score 2-3 on the Likert scale).
* Women between the ages of 40 and 65, inclusive, in the peri- or postmenopausal period.
* Women are able to understand and sign the informed consent after the nature of the study has been fully explained to them.

Exclusion Criteria:

* Pregnant or immediate postpartum patients (up to 40 days).
* Formal contraindication for the use of the product, such as hypersensitivity to any of the components of the study treatment.
* Use of any other experimental drug or device during the 30 days prior to screening.
* Use of topical antibiotics or antifungals applied vaginally in the two weeks prior to the initial visit.
* Use of contraceptives for vaginal application.
* Decompensated chronic diseases (diabetes, epilepsy, high blood pressure, etc.)
* Undiagnosed abnormal genital bleeding or presence of vaginal lesion.
* Active genitourinary infections at the time of inclusion or in the 15 days prior to inclusion in the study.
* Impossibility, at the discretion of the researcher, to comply with the requirements of the study, either due to follow-up problems, or due to their psychophysical characteristics.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women with vulvovaginal atrophy
Enrollment: 134 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-02 (Actual)

PRIMARY OUTCOMES:
Efficacy of Idracare® in the treatment of symptoms of vulvovaginal atrophy (VVA) | Through study completion, an average of 12 weeks
  To evaluate the efficacy of the Idracare® gel as a treatment for the symptoms of VVA, the percentage of women who present changes in dryness and / or dyspareunia has been established as the main variable.
Safety of Idracare® in the treatment of symptoms of vulvovaginal atrophy (VVA) measuring the incidence, nature and severity of adverse events (AE). | Through study completion, an average of 12 weeks
  To evaluate the safety of Idracare® gel, the incidence, nature and severity of adverse events (AE) will be studied.

SECONDARY OUTCOMES:
To evaluate the effect of Idracare® gel using Bachmann Vaginal Health Index (BVHI). | 4 and 12 weeks
  Effect of Idracare® gel will be evaluated on vaginal health status using Bachmann Vaginal Health Index (BVHI). It consists of 5 domains that evaluate different parameters (elasticity, fluids, pH, epithelial integrity and moisture) scoring each one of them independently, considering the maximum score as the best vaginal health status.
To evaluate the effect of Idracare® gel using vulvar health index (VHI). | 4 and 12 weeks
  Effect of Idracare® gel will be evaluated on vaginal health status using vulvar health index (VHI). It consists of 8 domains that evaluate different parameters: physiological state of the labia majora, labia minora, clitoris, urethra, coloration, elasticity / introitus, discomfort / pain and other findings) scoring each of them independently, considering the maximum score as the worse in vulvar health.
To evaluate the effect of Idracare® gel using vaginal pH | 4 and 12 weeks
  Effect of Idracare® gel will be evaluated on vaginal health status using vaginal pH changes. A lower pH compared to basal is considered an improvement on vaginal health status.
To evaluate the effect of Idracare® gel using maturation of vaginal epithelial cells. | 4 and 12 weeks
  Effect of Idracare® gel will be evaluated on vaginal health status using Maturation Index (MI). MI is the most commonly used index to assess hormonal status. It evaluates the percentage composition of the three large types of cells that make up the vaginal epithelium in the cytological samples obtained: parabasal, intermediate and superficial. It consists of selecting five fields at random (x 10 magnification) and counting 100 epithelial cells in each area, determining the percentage of superficial, intermediate and parabasal cells in each area. The result is expressed as% parabasal cells:% intermediate cells (navicular):% superficial cells.
To evaluate the effect of Idracare® gel using vaginal microbiota. | 4 and 12 weeks
  Effect of Idracare® gel will be evaluated on vaginal health status using vaginal Dysbiosis test. It consists of analyzing by means of real time polymerase chain reaction (real time PCR) different microorganisms that are part of the vaginal ecosystem such as Lactobacillus species (L. crispatus, L. jensenii, L. iners, L. gasseri ), Candida species, lactic acid microbiota (Atopobium, Gardnerella), non-lactic acid microbiota and pathogens.
The degree of satisfaction with the use of Idracare® | 4 and 12 weeks
  The degree of satisfaction with the use of Idracare® will be evaluated using a 7-point Likert-type scale, from 1 (satisfied) to 7 (not satisfied at all).
The tolerability of the treatment using a 5-point Likert-type scale | 4 and 12 weeks
  The tolerability of the treatment will be evaluated using a 5-point Likert-type scale, from 1 (no problem with the treatment) to 5 (I can't stand the treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Josep Combalia, MD, Study Director — Procare health Iberia; Fernando Losa, Doctor, Principal Investigator — Clínica Sagrada Familia; Santiago Palacios, Doctor, Principal Investigator — Instituto Palacios de Salud y Medicina de la Mujer
Locations (4):
- Spain (4):
  - Clínica Sagrada Familia, Barcelona
  - HM Gabinete Velázquez, Madrid
  - Instituto Palacios de Salud y Medicina de la Mujer, Madrid
  - HU Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
The study documentation will be shared after study completion
Supporting Information: Study Protocol, ICF, CSR